CLINICAL TRIAL: NCT02067572
Title: A Comparison of the Effectiveness of Normal Saline Mouthwash and Mouthwash Based on Tea Solution From Salvia Officinalis (SO) in Palliative Care. A Randomized Controlled Trial
Brief Title: A Randomized Controlled Trial Evaluating the Effectiveness of a Salvia-based Mouthwash in Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Salvia
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Terminal Illness; Xerostomia
Keywords: oral health; mouthwash; salvia; hospice; xerostomia; mouth sores
MeSH Terms: conditions — Xerostomia; Oral Ulcer

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salvia (Experimental): Salvia mouthwash used 4 times per day for 4 days
  Interventions: Other: Salvia mouthwash
- Saline (Active Comparator): Saline mouthwash used 4 times per day for 4 days.
  Interventions: Other: Saline mouthwash

INTERVENTIONS:
Other: Saline mouthwash
  Arms: Saline
Other: Salvia mouthwash
  Arms: Salvia

SUMMARY:
This study examines the effectiveness of an herbal mouthwash made from salvia in maintaining good oral health among patients in palliative care. It is hypothesized that using the mouthwash made from salvia will result in better oral health and more oral comfort than using with conventional normal saline mouthwash.

DETAILED DESCRIPTION:
The aim of this study is to examine the effectiveness of an herbal mouthwash made from salvia officinalis (SO) in maintaining good oral health among patients in palliative care. The study compares a mouthwash based on salvia tea solution with conventional normal saline mouthwash and addresses the following research questions:

1. Does the SO-based mouthwash provide a better treatment than conventional normal saline in maintaining good oral health in terminally ill patients?
2. Is there a difference in the individual perception of oral comfort in patients receiving SO versus patients receiving saline rinsing solution?

ELIGIBILITY:
Inclusion Criteria:

* Attending bedded unit at Hospice
* Over 18 years of age and able to provide written formal consent
* Diagnosed with advanced cancer
* Patient with positive response when asked if they experience oral discomfort or complications.

Exclusion Criteria:

* Estimated life expectancy prognosis of less than 2 weeks
* Significant cognitive impairment
* Current use of antifungal medication
* Currently receiving radiation therapy or chemotherapy
* Epileptic
* Diabetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2016-09-08 (Actual); Study Completion 2016-09-08 (Actual)

PRIMARY OUTCOMES:
Oral health (OMAS) | after 4 days of using mouthwash
  Oral Mucositis Assessment Scale (OMAS)
Patient's perception of oral comfort | after 4 days of using mouthwash
  Questions regarding oral discomfort and EORTC-OH17
Oral health (clinical evaluation) | after 4 days of using mouthwash
  Clinical evaluation by dentist

SECONDARY OUTCOMES:
General symptom experience | after 4 days of using mouthwash
  Edmonton Symptom Assessment System (ESAS)

CONTACTS AND LOCATIONS:
Overall Officials: Anners Lerdal, PhD, Principal Investigator — Lovisenberg Diakonale Hospital
Locations (1):
- Lovisenberg Hospice, Oslo, Norway

REFERENCES:
- [Derived] Monsen RE, Kristoffersen AK, Gay CL, Herlofson BB, Fjeld KG, Hove LH, Nordgarden H, Tollisen A, Lerdal A, Enersen M. Identification and susceptibility testing of oral candidiasis in advanced cancer patients. BMC Oral Health. 2023 Apr 18;23(1):223. doi: 10.1186/s12903-023-02950-y. PMID 37072843
- [Derived] Monsen RE, Herlofson BB, Gay C, Fjeld KG, Hove LH, Malterud KE, Saghaug E, Slaaen J, Sundal T, Tollisen A, Lerdal A. A mouth rinse based on a tea solution of Salvia officinalis for oral discomfort in palliative cancer care: a randomized controlled trial. Support Care Cancer. 2021 Sep;29(9):4997-5007. doi: 10.1007/s00520-021-06021-2. Epub 2021 Feb 14. PMID 33586003